CLINICAL TRIAL: NCT06142682
Title: Dexamethasone-Eluting Cochlear Implant Electrode (CIDEXEL): Pivotal Study
Brief Title: Dexamethasone Eluting Cochlear Implant: a Pivotal Study
Acronym: CDEX2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDEX2_MED-EL_CRD_2021_01
Record Dates: First submitted 2023-11-07; First posted 2023-11-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cochlear Implant
Keywords: cochlear implantation; CI; Dexamethasone
MeSH Terms: interventions — Cochlear Implants

STUDY DESIGN:
Intervention Model Description: The Cochlear Implant (CI) Mi1250 +FLEX28 DEX (CIDEXEL) is the Investigational Medical Device (IMD) under investigation. MED-EL CI systems consist of an implantable part (i.e. CIDEXEL), external components (i.e. technically compatible audio/speech processor and its accessories) and software that controls and powers the implant. The IMD CIDEXEL will be the implantable part of this new MED-EL CI System and shall only be used together with technically compatible MED-EL external components.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIDEXEL (Experimental): MED-EL Cochlear Implant Mi1250 +FLEX28 DEX (CIDEXEL)
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — cochlear implantation with dexamethasone eluting electrode

SUMMARY:
The newly developed MED-EL Cochlear Implant Mi1250 +FLEX28 DEX (CIDEXEL) incorporates the anti-inflammatory agent dexamethasone (DEX) into the electrode array. The passive elution of DEX during the post-implantation period has the purpose of counteracting the increase of the post-operative impedance induced by the insertion trauma.

The aim of this clinical investigation is to obtain confirmatory data concerning safety and performances of the investigational device in the clinical population.

DETAILED DESCRIPTION:
The Cochlear Implant Mi1250 +FLEX28 DEX (CIDEXEL) is the Investigational Medical Device (IMD) under investigation. MED-EL CI systems consist of an implantable part (i.e. CIDEXEL), external components (i.e. technically compatible audio/speech processor and its accessories) and software that controls and powers the implant. The IMD CIDEXEL will be the implantable part of this new MED-EL CI System and shall only be used together with technically compatible MED-EL external components.

None of the components mentioned above incorporates, as an integral part transplants or tissues or cells of human or animal origin. No products incorporating or derived from tissues or cells of human or animal origin were used during its manufacturing.

• Primary Objective

The primary objective of this clinical investigation is to confirm the clinical performance of the CIDEXEL by comparing Speech intelligibility results measured pre-operatively to those measured at the 6-months follow-up.

For this clinical investigation to be successful, mean speech test results at the 6-months visit shall be superior to the mean speech test results obtained pre-operatively. (Monosyllables)

• Secondary Objectives

The secondary objectives of this clinical investigation are to measure:

* Impedance Field Telemetry (IFT) values and derived measures
* Fitting Maps reiteration appraisal
* Electrically evoked Compound Action Potential (eCAP) and derived measures
* Unaided audiograms obtained pre- and post-operatively
* Hearing Preservation (HP) %
* The improvement in generic quality of life (measured by the Health Utilities Index (HUI2&3)) pre- to the 6-months visit
* The improvement in disease specific quality of life (measured by the Nijmegen Cochlear Implant Questionnaire (NCIQ)) pre- to the 6-months visit
* Surgical Usability and satisfaction (Ad Hoc questionnaire for the surgeons )
* Sentence test in noise results across the tested intervals (OlSa)
* Speech, spatial and quality of hearing across the tested intervals (Speech, Spatial and Qualities of hearing scale (SSQ12))
* Sound quality over time (Hearing Implant Sound Quality Index (HISQUI))
* Wearing time (data Logging)
* Safety Objective

The purpose of this clinical investigation is to establish and verify the clinical safety of the CIDEXEL. To confirm the safety profile of the device which will be evaluated through the analysis of adverse events during the follow-up period. For the study to be considered a success, the results of the adverse event analysis shall never cause an unbalanced risk vs. benefit assessment biased towards the former.

ELIGIBILITY:
Inclusion Criteria:

Minimum age of eighteen (18) years at time of enrolment.

* Hearing loss on the ipsilateral ear (see Figure 8 for the specific audiological criteria).
* A functional auditory nerve in the ear to be implanted.
* Subjects reporting to having used an optimally fit hearing aids for a minimum of three months before the decision that a cochlear implant is the preferential option.
* Cochlea anatomy compatible with the insertion of a FLEX28 electrode array.
* Compatibility with a soft surgery approach as per clinical practice at the site.
* Post-lingual hearing impairment.
* Subject fulfilling indication criteria for a CI according to the local professional standards, as reported by the implanting surgeon.
* General health condition, psychological and emotional condition deemed compatible with the treatment and tests performed in this study and realistic expectations, as deemed appropriate by the implanting surgeon.
* Signed and dated informed consent before the start of any study-specific procedure.

Exclusion Criteria:

* Lack of compliance with any inclusion criterion.
* Previously having received a cochlear implant on the ear chosen for placing the IMD.
* Evidence of ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array or might cause increased risk of infection (e.g. dysplastic cochlea), as confirmed by medical examination and/or as per CT/MRT.
* Evidence of anatomic abnormalities that would prevent appropriate placement of the stimulator housing in the bone of the skull.
* Known allergic reaction or intolerance to the materials used in the implant (including medical grade silicone, platinum, iridium, parylene c, DEX).
* Known absence of cochlear development or if the cause of deafness is non-functionality of the auditory nerve and/or the upper auditory pathway.
* Evidence of active external or middle ear infection or history of recurrent middle ear infection in the ear to be implanted.
* Evidence of perforated tympanic membrane in the ear to be implanted.
* Patient reporting immunosuppressive therapy or corticosteroids therapy in the 4 weeks before enrolment.
* Evidence of concomitant use of medicinal substances that, in the opinion of the investigator, could alter the therapeutic efficacy of dexamethasone.
* Unwillingness or inability of the candidate to comply with all investigational requirements.
* Evidence of medical contraindications to surgery of the middle and inner ear and anaesthesia.
* Additional disabilities that would prevent or restrict participation in the audiological and medical evaluations required of the clinical investigation.
* Subject not capable of giving consent.
* Individual subjected to court-ordered or government-authorized deprivation of liberty as defined by § 27 MPDG.
* Evidence of Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean/median speech perception outcome as % correct of speech test in quiet from prior to implantation to the 6-months follow-up with the CIDEXEL | 6 months visit
  Speech intelligibility results measured pre-operatively to those measured at the 6-months follow-up.

SECONDARY OUTCOMES:
IFT | 6 months visit
  Impedance Field Telemetry data in kOhm per channel
eCAP | 6 months visit
  Interphase Gap analysis per electrode in charge units
Hearing Preservation % | 6 months visit
  Hearing preservation calculated according to the HEARRING HP scale in %
HUI 3 (Health Utility Index) | 6 months visit
  Questionnaire outcomes (scale where dead = 0.00 and perfect health = 1.00)
NCIQ (Nijmegen Cochlear Implant Questionnaire) | 6 months visit
  Questionnaire outcomes (Physical, Psychological and Social functioning) score 0-100
ad Hoc Surgical questionnaire | 6 months visit
  Questionnaire outcomes descriptively apprised
OlSa | 6 months visit
  Speech Intelligibility testing outcomes in dB
SSQ12 (Speech Spatial Quality of hearing) | 6 months visit
  Questionnaire outcomes Scores 0-10
HISQUI (Hearing Implant Sound Quality Index) | 6 months visit
  Questionnaire outcome: very poor sound quality < 30, poor sound quality 30 - 60, moderate sound quality 60 - 90, good sound quality 90 - 110, very good sound quality 110 - 133
Wearing time | 6 months visit
  Audio processor wearing time in min

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Plontke, Prof. Dr., Principal Investigator — Martin-Luther-Universität Halle-Wittenberg, Universitätsklinik und Poliklinik für Hals-Nasen-OhrenHeilkunde, Kopf- und Hals-Chirurgie
Locations (7):
- Germany (7):
  - HNO-Klinik der Ruhr-Universität Bochum, Bochum
  - Klinik und Poliklinik für Hals-, Nasen- und Ohrenheilkunde, Dresden
  - Universitätsklinikum Frankfurt Klinik für HNO-Heilkunde, Frankfurt
  - Martin-Luther-Universität Halle-Wittenberg, Universitätsklinik und Poliklinik für Hals-Nasen-OhrenHeilkunde, Kopf- und Hals-Chirurgie, Halle
  - HNO-Klinik der Medizinischen Hochschule Hannover, Hanover
  - Universitätsklinik für Hals-, Nasen- und Ohrenheilkunde, Tübingen
  - Klinik und Poliklinik für Hals-, Nasen- und Ohrenkrankheiten, plastische und ästhetische Operationen. Die Universitäts-HNO-Klinik Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No